CLINICAL TRIAL: NCT01763138
Title: Effect of Educational Intervention in Mothers for Prevention of Caries in Their Children, A Randomized Controlled Trial
Brief Title: Effect of Educational Intervention in Mothers for Prevention of Caries in Their Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Collaborators: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Responsible Party: Principal Investigator, Dr Fatima Ishfaq, Dr. Fatima Ishfaq, University of the Punjab
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: fatima ishfaq
Record Dates: First submitted 2013-01-06; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Health Education, Dental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pamphlet and reminder (Other): pictorial oral health pamphlet comprising of instructions on child's oral hygiene and feeding practices and a oral health education reminder phone call after a period of one month.
  Interventions: Behavioral: oral health education; Behavioral: reminder phone call
- pamphlet only (Other): oral health education pictorial pamphlet would be provided to mothers however there will be no reminder phone calls.
  Interventions: Behavioral: oral health education
- control (No Intervention): no oral health education or reminder phone calls will be provided to mothers.

INTERVENTIONS:
Behavioral: oral health education — oral health education in the form of a pictorial pamphlet.
  Arms: pamphlet and reminder; pamphlet only
Behavioral: reminder phone call — a reminder phone call on oral health instructions would be given to mothers after every one month over a period of three months.
  Arms: pamphlet and reminder

SUMMARY:
The purpose of this study is to determine the effect of an educational intervention on mothers knowledge, attitudes and practices for preventing childhood caries.

DETAILED DESCRIPTION:
Health education is being used as a key preventive tool in the prevention of chronic diseases such as heart disease, cancer, obesity, mental illness, neurological disturbances as well as dental diseases.

Amongst the dental diseases, dental caries is a high prevalence chronic childhood disease having long term growth and developmental implications . A number of educational programs have been utilized to decrease its prevalence especially in disadvantaged communities.

Dental caries is a complex interplay of a number of risk factors such as demographic (socioeconomic status, race, etc.) behavioral, dietary and cultural factors. Among the dietary intake, the most significant risk factor has been a high frequency intake of sugary foods and drinks.Patterns of sugar intake are established early in life and sugar intake increases in the first two years of life.

Early feeding practices and lack of oral hygiene maintenance have been identified as risk factors for caries in subsequent years. Maternal education can prove to be protective against dental caries by way of child's dietary practices.

Research has also indicated a reduction in prevalence of caries in children whose parents were previously participants of an oral health educational program.

Educating mothers about oral hygiene and feeding practices before the child transitions from exclusive milk diet to a variety of foods in an important time to exert a positive influence on dietary intake of child and overall oral health.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of 9-15 months old attending the vaccination clinic who consented to be a part of the study

Exclusion Criteria:

* Mothers with severely ill children or children suffering from a co-morbid disease.

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
improvement in child's oral hygiene | 3 months
  Increase in the frequency of tooth brushing, use of a proper oral hygiene aid would indicate an improvement in the child's oral hygiene as reported by the mother after a three month follow up period.

SECONDARY OUTCOMES:
reduction in sugar intake | 3 months
  A reduction in child's sugar intake would be assessed through the followup structured questionnaire as reduced frequency of sugary snacking and a reduction in night time feeding practices.

OTHER OUTCOMES:
Improvement in Mothers knowledge and attitudes regarding their child's oral health | 3 months
  An improvement in mother's knowledge and attitudes regarding their child's oral health would be assessed through the part of the questionnaire comprising of questions on fluoride, importance of milk teeth, prevention of caries etc

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Ishfaq, BDS, Principal Investigator — Sheikh Zayed Federal Postgraduate Medical Institute
Locations (1):
- Children Hospital and Institute of Child Health, Lahore, Punjab Province, Pakistan